CLINICAL TRIAL: NCT03000231
Title: Circadian Function and Cardio-metabolic Risk in Adrenal Insufficiency: a Case Control Study
Brief Title: Circadian Function and Cardio-metabolic Risk in Adrenal Insufficiency
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1484
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls: Matched by age, race, gender and BMI to adrenal insufficiency subjects
- Adrenal Insufficiency Patients: Eligible patients will have either primary adrenal insufficiency or secondary adrenal insufficiency and will be age 18 and older.

SUMMARY:
The purpose of this study is to compare cardio-metabolic risk, glucose tolerance, and night time blood pressure between healthy control subjects and patients with adrenal insufficiency. No intervention will be administered and the study is observational only.

DETAILED DESCRIPTION:
We propose to use a case control design to test the main hypothesis that as compared to healthy control subjects matched for sex, age, adiposity and race/ethnicity, patients with adrenal insufficiency, whether primary or secondary, have disturbances of the circadian system that are associated with high day to day variability of sleep time as well as elevated markers of cardio-metabolic risk, including abnormal oral glucose tolerance and reduced nocturnal blood pressure dipping.

A secondary hypothesis of the study is that adrenal insufficiency patients on a replacement regimen (as part of their standard of care ongoing treatment) that results in daytime cortisol profiles approximating the normal diurnal variation will have better cardio-metabolic function than adrenal insufficiency patients who have grossly abnormal cortisol profiles.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary adrenal insufficiency, Healthy matched controls, acute or unstable health conditions age 18 or older

Exclusion Criteria:

* Diabetes, Tertiary adrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary Adrenal Insufficiency age 18 and older and healthy matched control subjects
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
day to day variability of sleep timing over 1 week of recording | day 1 to day 7
  On each day, the midpoint (time in hours and minutes) of the sleep period will be calculated and the variability over 1 week will be quantified by the standard deviation

SECONDARY OUTCOMES:
nocturnal blood pressure dipping | day 8 to 9
  a 24-h recording of blood pressure will be conducted in the laboratory with concurrent sleep recording. Dipping will be calculated as the difference between the daytime mean and the nighttime mean
oral glucose tolerance | day 11 to 12
  A 3-h 75g oral glucose tolerance test will be performed in the laboratory after an overnight fast. Glucose tolerance will be quantified by the total area under the glucose curve over the 3-hour period of sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No